CLINICAL TRIAL: NCT00413374
Title: Once Daily Enoxaparin for Outpatient Treatment of Acute Deep Venous Thrombosis and/or Pulmonary Embolism
Brief Title: Once Daily Enoxaparin for Outpatient Treatment of Acute DVT and/or Pulmonary Embolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Samuel Z.Goldhaber, MD, Director, VTE Research Group, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-000082
Record Dates: First submitted 2006-12-15; First posted 2006-12-19 (Estimated); Results first posted 2012-04-30 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Lovenox; Enoxaparin; Prophylaxis; Pulmonary Embolism; Acute Deep Vein Thrombosis; Venous Thrombosis; Thrombosis; Anticoagulation
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enoxaparin (Other)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Patient takes 1.5 mg per kilogram, once daily, subcutaneous injections until INR is therapeutic, then medication is stopped.
  Other Names: Lovenox

SUMMARY:
To investigate the efficacy and safety of once daily enoxaparin as a "bridge" to warfarin for the outpatient treatment of acute deep venous thrombosis or pulmonary embolism.

DETAILED DESCRIPTION:
Background and Significance:

Low molecular weight heparin (LMWH) as a "bridge" to warfarin has become the standard of care for outpatient treatment of acute deep venous thrombosis (DVT). LMWH is also often prescribed as a "bridge" to warfarin for patients with acute pulmonary embolism (PE). In the United States, the FDA has approved enoxaparin only for twice daily dosing in outpatient treatment of acute DVT. The FDA has also approved enoxaparin for treatment of DVT with or without PE, but the FDA has not approved enoxaparin for the treatment of PE without DVT. The FDA has also not approved once daily enoxaparin for any DVT or PE treatment indication for outpatients.

Once daily dosing of enoxaparin in outpatients with DVT alone, DVT with PE, or PE without DVT will halve the number of required injections, facilitate outpatient treatment, and reduce health care costs. For example, visiting nurses will make one visit daily instead of two visits daily for those patients who are unable self-inject and for those patients who lack family or friends to inject LMWH.

Merli et al randomized 900 hospitalized venous thromboembolism (VTE) patients with acute DVT or PE to one of three treatment groups: 1) continuous infusion of unfractionated heparin (UFH), 2) once daily enoxaparin 1.5mg/kg, or 3) twice daily enoxaparin 1mg/kg. All study patients were inpatients. None were outpatients. They received once or twice daily enoxaparin or UFH for at least five days and were "bridged" to warfarin. Patients were followed for three months. Primary endpoints were recurrent DVT or PE. There were no significant differences in recurrent DVT or PE among the 3 treatment groups. There were 12 recurrent VTE events in the UFH group, 13 in the once daily enoxaparin group, and 9 in the twice daily enoxaparin group.

The frequency of major hemorrhage did not differ among the three treatment groups. Major hemorrhage occurred in 6 of 290 patients (2.1%) in the UFH group, 5 of 298 patients (1.7%) in the once daily enoxaparin group, and 4 of 312 patients (1.3%) in the twice daily enoxaparin group.

Merli et al showed that once daily enoxaparin was as effective and safe as twice daily enoxaparin. But this study was done only among hospitalized patients with acute DVT or PE. Treatment results in hospitalized patients do not necessarily apply to the outpatient population. Therefore, the FDA has not approved outpatient DVT or PE treatment with once daily enoxaparin.

The BWH Venous Thromboembolism Research Group has an outstanding track record for investigator initiated trials. We have recently completed 2 investigator initiated trials with enoxaparin for the treatment of PE. One trial was published in Thrombosis and Haemostasis and the other is accepted for publication in Vascular Medicine.

Clinically stable PE patients with normal right ventricular size and function as assessed by echocardiogram or chest CT scan are at very low risk of adverse clinical events. Either imaging test is excellent for acquiring the information we need to document normal RV size and function. These clinically stable PE patients with negative biomarkers (troponin) and normal right ventricular function can be safely treated as outpatients.

Therefore, we wish to include in this trial clinically stable patients with acute PE who have normal right ventricular size on chest CT in addition to patients with acute DVT. Chest CT with a 4 chamber view with RVD/LVD measurement will be performed in all cases by a radiologist with experience in this technique to confirm normal RV size on all PE patients.

In this investigator initiated trial, we will conduct a feasibility study with once daily enoxaparin as a "bridge" to warfarin for outpatient treatment of acute DVT or PE.

Subject selection:

Physicians caring for DVT and PE patients in the noninvasive vascular lab, Emergency Department, primary care office, and inpatient care units at Brigham and Women's Hospital often summon our Group for consultation. Our Group will under these circumstances describe this protocol. If the referring physician and the patient agrees, these patients will be approached for enrollment by physician investigators from the research team.

We will study 40 patients with symptomatic DVT or PE confirmed by ultrasound or chest computed tomography respectively and treat them with once daily enoxaparin as a bridge to warfarin. In this case-control series, we will match 2 historical controls by age and gender to every case. Controls who received twice daily enoxaparin as a "bridge" to warfarin for acute venous thromboembolism will be matched from a retrospective study of previously hospitalized patients. Additional characteristics of matched control group will include: prior DVT or PE, cancer, heart disease, and pulmonary disease.

All patients enrolled in the study will receive enoxaparin 1.5mg/kg/day as a bridge to warfarin, using at least 4 outpatient doses of enoxaparin and overlapping enoxaparin and warfarin for at least 4 days.

Study Procedures:

Enrollment: Eligible patients with confirmed DVT and/or PE who are stable for outpatient treatment will be approached for enrollment.

Following enrollment, patients will be started on enoxaparin 1.5mg/kg/day as a bridge to warfarin. Patients will receive overlapping once daily enoxaparin and warfarin for at least 4 days.

After enrollment, patients will be started on warfarin 7.5 mg daily. Initial INR will be checked on day 3 after starting warfarin. Thereafter, INR will be checked daily from day 4 to day 7 and until INR is ≥ 2.0 for 2 consecutive days. Enoxaparin will be discontinued after a minimum of 4 days and after 2 consecutive values ≥ 2.0. Once enoxaparin is discontinued patients will continue oral warfarin alone. All INR tests can be done at any hospital, including Brigham and Women's, or at a lab that is closer to patient's home.

Study investigators will perform anticoagulation management after discharge for 30 days; with an initial office follow-up visit between days 7 and 13 and a final office visit between days 27 and 33. This will include clinical assessment, and blood testing of renal function and international normalized ratio (INR). Each study visit will take up to 1 hour. Each blood test will require 5 ml of patient's blood.

At the conclusion of the 30-day trial, responsibility for anticoagulation, including the decision about its duration, will revert to the Primary Care Physician.

Biostatistical Analysis:

The sample size of 40 patients serves to assess the feasibility and safety of once daily enoxaparin therapy as a bridge to warfarin for outpatient treatment of acute DVT and/or PE.

A composite endpoint of death, recurrent venous thromboembolism, and major hemorrhage will be assessed at 30 days. Comparisons are made on an intention-to-treat basis. Separate analyses will also be performed on each individual endpoint.

The statistical analysis plan will include specific exploratory subgroup analyses: DVT without PE, PE without DVT, and combined DVT plus PE.

The statistical analysis will be by "intention to treat." In other words, once a patient is recruited, that patient will be analyzed regardless of protocol violations and regardless of missing data. No patient will be excluded from the analyses because of protocol violations, missing data, or any other reason.

Chi-squared testing will be used for statistical analysis. For cells with 5 or fewer patients, the Fisher's Exact Test will be used.

Efficacy and safety will be statistically evaluated in a composite endpoint. This composite endpoint will include: Death, recurrent venous thromboembolism, and major hemorrhage at 30 days. Separate analyses will also be performed on each individual endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic acute deep venous thrombosis and/or pulmonary embolism confirmed by venous ultrasound and/or CT scan.
2. Pulmonary embolism patients with normal right ventricular size on chest CT scan.
3. Age greater than 18 years
4. Anticipated discharge within 72 hours of admission
5. Written informed consent

Exclusion Criteria:

1. Pregnancy or intend to become pregnant
2. Patients requiring ongoing hospitalization > 72 hours
3. Hypersensitivity to heparin, pork products or enoxaparin
4. Creatinine > 2.0 mg/dl
5. Recurrent DVT and/or PE with oral anticoagulation
6. Surgery or medical procedure planned during the study that may pose a significant bleeding risk
7. Prior history of heparin-induced thrombocytopenia
8. Inability to participate for follow up appointments and study visits
9. Life expectancy < 30 days
10. High risk of bleeding:

    1. Active major bleeding within 30 days by GUSTO criteria
    2. History of intracranial bleeding
    3. Major surgery or trauma within 10 days
    4. Head injury requiring hospitalization within 1 year
    5. Intracranial tumor
    6. Neurosurgery or non-cataract ophthalmologic surgery within 1 month
    7. Thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z. Goldhaber, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Merli G, Spiro TE, Olsson CG, Abildgaard U, Davidson BL, Eldor A, Elias D, Grigg A, Musset D, Rodgers GM, Trowbridge AA, Yusen RD, Zawilska K; Enoxaparin Clinical Trial Group. Subcutaneous enoxaparin once or twice daily compared with intravenous unfractionated heparin for treatment of venous thromboembolic disease. Ann Intern Med. 2001 Feb 6;134(3):191-202. doi: 10.7326/0003-4819-134-3-200102060-00009. PMID 11177331
- [Background] Beckman JA, Dunn K, Sasahara AA, Goldhaber SZ. Enoxaparin monotherapy without oral anticoagulation to treat acute symptomatic pulmonary embolism. Thromb Haemost. 2003 Jun;89(6):953-8. PMID 12783106
- [Background] Kucher N, Quiroz R, McKean S, Sasahara AA, Goldhaber SZ. Extended enoxaparin monotherapy for acute symptomatic pulmonary embolism. Vasc Med. 2005 Nov;10(4):251-6. doi: 10.1191/1358863x05vm634oa. PMID 16444853
- [Background] Kucher N, Rossi E, De Rosa M, Goldhaber SZ. Prognostic role of echocardiography among patients with acute pulmonary embolism and a systolic arterial pressure of 90 mm Hg or higher. Arch Intern Med. 2005 Aug 8-22;165(15):1777-81. doi: 10.1001/archinte.165.15.1777. PMID 16087827
- [Background] Schoepf UJ, Kucher N, Kipfmueller F, Quiroz R, Costello P, Goldhaber SZ. Right ventricular enlargement on chest computed tomography: a predictor of early death in acute pulmonary embolism. Circulation. 2004 Nov 16;110(20):3276-80. doi: 10.1161/01.CIR.0000147612.59751.4C. Epub 2004 Nov 8. PMID 15533868
- See also: North American Thrombosis Forum — http://www.NATFonline.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in September 2006 and was completed in March 2008. Of 473 patients screened, 40 were enrolled.
  Patients with newly diagnosed acute DVT or PE were screened in the Emergency Department or Vascular Laboratory at Brigham and Women's Hospital.
Units Other Than Participants: patients
Groups:
- Enoxaparin 1.5 mg/kg Daily: the cases were started on 1.5 mg/kg once daily enoxaparin as a bridge to warfarin.
- Enoxaparin 1 mg/kg Twice Daily: The controls had been treated with enoxaparin 1 mg/kg twice daily as a ''bridge'' to warfarin.
  These are historical controls.
  Two previously treated controls were matched for each case. Controls were matched by age (+10 years), gender, and location of VTE. The controls had been treated with enoxaparin 1 mg/kg twice daily as a ''bridge'' to warfarin.
Period: Overall Study
Arm/Group | Enoxaparin 1.5 mg/kg Daily | Enoxaparin 1 mg/kg Twice Daily
Started | 40; 40 patients | 80; 80 patients
Completed | 34; 34 patients | 80; 80 patients
Not Completed | 6; 6 patients | 0; 0 patients
Not completed — Ineligible due to screening criteria. | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Surgery | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enoxaparin 1.5 mg/kg Daily | Enoxaparin 1 mg/kg Twice Daily | Total
Number analyzed (Participants) | 40 | 80 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 75 | 110
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.95 (16.2) | 48.53 (15.3) | 48 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 42 | 63
  Male | 19 | 38 | 57
Region of Enrollment [Number; unit: participants]
  United States | 40 | 80 | 120

OUTCOME MEASURES:

1. Primary Outcome: Major Bleeding Complication
Description: Major bleeding complication as defined as spinal, retroperitoneal, or intracranial bleeding; drop in hemoglobin ≥2g/dl or transfusion ≥2U or surgical or medical intervention, death related to bleeding.
Time Frame: 30 Days
Measure: Number; unit: participants
Groups:
- Enoxaparin 1.5 mg/kg Daily: Study participants receiving Enoxaparin once daily who developed a major bleeding complication within 30 days.
Arm/Group | Enoxaparin 1.5 mg/kg Daily | Enoxaparin 1 mg/kg Twice Daily
Number analyzed (Participants) | 40 | 80
participants | 0 | 3

2. Primary Outcome: Recurrent VTE
Description: Major clotting complication (recurrent VTE) as defined as recurrent acute pulmonary embolism confirmed on chest CT or recurrent deep vein thrombosis in the contralateral extremity confirmed with venous ultrasound or CT scan while on once daily enoxaparin therapy.
Time Frame: 30 Days
Measure: Number; unit: participants
Groups:
- Enoxaparin 1.5 mg/kg Daily: Participants receiving Enoxaparin once daily who developed a VTE (either a DVT or PE) within 30 days.
Arm/Group | Enoxaparin 1.5 mg/kg Daily | Enoxaparin 1 mg/kg Twice Daily
Number analyzed (Participants) | 40 | 80
participants | 1 | 3

3. Primary Outcome: Death
Description: All-cause mortality
Time Frame: 30 Days
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Groups:
- Enoxaparin 1.5 mg/kg Once Daily: the cases were started on 1.5 mg/kg once daily enoxaparin as a bridge to warfarin
- Enoxaparin 1 mg/kg Twice Daily: The controls had been treated with enoxaparin 1 mg/kg twice daily as a ''bridge'' to warfarin.
Arm/Group | Enoxaparin 1.5 mg/kg Once Daily | Enoxaparin 1 mg/kg Twice Daily
Number analyzed (Participants) | 40 | 80
Participants | 0 | 0

ADVERSE EVENTS:
Groups:
- Enoxaparin 1.5 mg/kg Daily: Recieved low molecular weight heparin (LMWH) as a "bridge" to warfarin
Arm/Group | Enoxaparin 1.5 mg/kg Daily | Enoxaparin 1 mg/kg Twice Daily
Serious Adverse Events (participants affected / at risk) | 1/40 | 3/80
Other Adverse Events (participants affected / at risk) | 0/40 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enoxaparin 1.5 mg/kg Daily (N=40) | Enoxaparin 1 mg/kg Twice Daily (N=80)
Recurrent VTE (Cardiac disorders) | 1 (1) | 3 (3) — The sole recurrent VTE in the once daily enoxaparin group was caused by heparin-induced thrombocytopenia with thrombosis in a patient who had been recently exposed to UFH.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No